CLINICAL TRIAL: NCT05467085
Title: Imaging-Guided Low Intensity Focused Ultrasound (LIFU) Neuromodulation of Ventral Striatum in Obsessive-Compulsive Disorder (OCD)
Brief Title: Imaging-Guided Low Intensity Focused Ultrasound (LIFU)
Acronym: LIFU
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Massachusetts General Hospital (Other); M.D. Anderson Cancer Center (Other)
Responsible Party: Principal Investigator, Wayne Goodman MD, Chair/Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-51465
Record Dates: First submitted 2022-06-21; First posted 2022-07-20 (Actual); Last update posted 2025-08-18 (Actual); Status verified 2025-08

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: OCD; LIFU; Low Intensity Focused Ultrasound
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Intervention Model Description: This open-label early feasibility study will be conducted in 20 subjects with OCD across two centers, Baylor College of Medicine (BCM)and Massachusetts General Hospital (MGH).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- LIFU in OCD group (Experimental): Each subject will receive 3 LIFU sessions epr week for two weeks (6 total image-guided treatments).
  A total of 20 sonications will be administered to one side of the head, with a derated (based on FDA standard of 0.3 dB/cm-MHz) spatial-peak temporal-average intensity (i.e., Ispta) of approximately 720mW/cm2, each lasting 30 s, separated by 30 s pause intervals. Thus, total duration of sonication will be 10 minutes, the same as used in our study of VS LIFU in healthy subjects. Sonication will be administered within a 3T Siemens Prisma scanner. During sonication, we will use the 20-channel head coil as the 32-or 64-channel coil does not allow enough space to fit the transducer.
  In summary, the entire sequence of 20 sonications, each lasting 30s, separated by 30s pause intervals, will be administered over 20 minutes for a total duration of sonication equal to 10 minutes.
  Interventions: Device: BX Pulsar 1002

INTERVENTIONS:
Device: BX Pulsar 1002 — Imaging-Guided Low Intensity Focused Ultrasound Pulsation (LIFU) device
  Other Names: Low Intensity Focused Ultrasound Pulsation (LIFUP)

SUMMARY:
This research study is to investigate the safety, feasibility, and possible therapeutic benefits of a technology called Low Intensity Focused Ultrasound (LIFU) in patients with obsessive- compulsive disorder (OCD). The device used in this study transmits high frequency sound waves to a particular region of the brain called the Ventral Striatum (VS). LIFU is a non-invasive form of stimulation, which can be used to stimulate deep regions of the brain. In this study, the investigators will administer LIFU to activate the VS area of the brain while also observing this brain stimulation with an MRI machine. Other aims of this study include learning more about the patterns of brain activity associated with OCD and seeing if brain activity changes as symptoms of OCD change over time during the two weeks of LIFU stimulation. Participants in this study will be asked to perform computer administered behavioral tasks -- similar to simple computer games -- to examine whether certain features of OCD (e.g., avoidance of feared triggers) change over the course of LIFU stimulation.

The treatment phase of this research study is expected to last two weeks with three weekly (total of 6) treatment sessions all carried at the MRI brain imaging center at Baylor College of Medicine. There will be at least one additional screening visit before treatment starts and a series of follow up visits over a six-month period.

DETAILED DESCRIPTION:
The current project will investigate a novel neurostimulation approach, low intensity focused ultrasound (LIFU), which combines non-invasiveness and a sharp spatial focus in deep brain regions. This open-label early feasibility study will be conducted in 20 subjects with OCD across two centers, Baylor College of Medicine (BCM) and Massachusetts General Hospital (MGH). Eligible subjects must have failed ERP and at least two trials of SRIs.

The study will use an MR-compatible Brainsonix (Pulsar 1002) transcranial device containing a single-element, air-backed, spherical section LIFU transducer with a diameter of 61mm and focal depth of either 65mm or 80mm, operating at a fundamental frequency of 650kHz. The selection of either a 65mm or 80mm transducer (as well as 0 or 5 gel pad) will depend upon the individual patient's head size/brain anatomy to optimally target the VS. The transducer is mounted in a plastic head holder and ultrasonic gel pad. LIFU will be administered in the Siemens Prisma 3T MR scanner to enable precise targeting of the ventral striatum (VS).

Each subject will receive 3 LIFUP sessions per week for two weeks (total=6 image-guided treatments). LIFU intensity will be at or below FDA safety limit of 720 mW/cm^2 Ispta, which resulted in an IRB/FDA determination of Non-Significant Risk (NSR) in our study of LIFU targeting the VS in healthy subjects. Outcome measures include safety (e.g., vital signs, adverse event reporting, tolerability, etc.), standardized symptom scales (e.g., change in YBOCS from baseline to assess OCD severity) as well as surrogate measures (e.g., behavioral tasks that assess constructs central to OCD). Subjects will be assessed clinically weekly for 8 weeks and then monthly for total of 6 months. Resting-state fMRI will be performed at baseline and at the end of the two-week study to assess changes in functional connectivity induced by LIFU treatment.

A total of 20 sonications will be administered to one side of the head, with a derated (based on FDA standard of 0.3 dB/cm-MHz) spatial-peak temporal-average intensity (i.e., Ispta) of approximately 720mW/cm2, each lasting 30 s, separated by 30 s pause intervals. Thus, total duration of sonication will be 10 minutes, the same as used in our study of VS LIFU in healthy subjects. Sonication will be administered within a 3T Siemens Prisma scanner. During sonication, the investigators will use the 20-channel head coil as the 32-or 64-channel coil does not allow enough space to fit the transducer.

Once the patient is brought to the MR suite, the investigators will acquire baseline resting-state BOLD MRI without the transducer in the coil. Then, the participant is taken out of the scanner, and the transducer is manually placed and secured to one side of the patient's head, over the temporal bone thinning. Using a lower resolution/faster acquisition T1 MPRAGE in a 3D MPR view, the investigators will navigate to the center of the transducer in one of the windows (sagittal). Then in both the coronal and axial views, the investigators will move the axes so that one is parallel to the face of the transducer, and then the other axis is positioned perpendicularly to it. The investigators will then trace the trajectory of both perpendicular axes to the appropriate focal depth. The investigators will then determine if the investigators are on target or not, estimate how much to adjust if necessary, pull the subject out, adjust as necessary, and repeat the process. Once the investigators are satisfied that the positioning is satisfactory, the investigators will proceed with a pilot stimulation straddled by a pair of baseline and post-stimulation ASL perfusion MRI scans and BOLD fMRI with concurrent LIFU stimulation. Then, the subject will once again be removed from the scanner, the transducer will be removed, and post-stimulation resting-state fMRI, high resolution anatomical scans (for image registration) and diffusion MRI will be collected. The LIFUP installation includes a 10 MHz low-pass filter to limit RF noise interference.

In summary, the entire sequence of 20 sonications, each lasting 30s, separated by 30s pause intervals, will be administered over 20 minutes for a total duration of sonication equal to 10 minutes. A physician will remain in the MR suite during the entire time. The subject will be given a squeeze ball switch for use in emergency, and the investigators will communicate with the subject regularly in between scans. Subject will remain in clinic for at least 30 minutes following the treatment. Vital signs, adverse events and self-report measures of mood and anxiety will be recorded.

Massachusetts General Hospital will obtain local IRB approval for their portion of this study

ELIGIBILITY:
Inclusion Criteria:

* 1. Outpatients, males and females, 21-55 years of age.
* 2. Principal diagnosis of OCD according to the DSM-5 with duration of ≥2 years.
* 3. Subjects with at least moderate OCD, defined by Yale-Brown Obsessive Compulsive Scale (YBOCS) (27) score of >19.
* 4. Had trials of at least two SSRIs or one SSRI and clomipramine.

  1. Treatment failure/non-response: As per the MGH-TRQ-OCD, minimal or no meaningful clinical benefit despite an adequate dose and duration of treatment;
  2. Adequate duration: At least 8 weeks of treatment with SSRI or clomipramine
  3. Adequate dose: Defined by the USPI labeling
* 5. If on medication, must be maintained on SRI medications at a stable therapeutic dosage for at least 2 months prior to study entry and for the duration of the trial.
* 6. If subjects are currently undergoing Exposure and Response Prevention (ERP) treatment, they must be in the maintenance stage with stable ERP "dosing" for at least 2 months.
* 7. Willing and able to adhere to the study schedule, which requires 6 sonication/scan visits over two weeks and follow up visits for up to 6 months.

Exclusion Criteria:

* 1.Subjects will be excluded with a history of more than four (4) previous failed treatment trials of SSRIs or clomipramine (not including any current medication trial) given for an adequate duration at an adequate dose.
* 2. Experimental therapy, either medication or device, within past 30 days.
* 3. TMS in last 30 days.
* 4. Present suicidal risk as assessed by the investigator using the Columbia Suicide Severity Rating Scale (28) or a history of attempted suicide in the past year.
* 5. History of epilepsy or seizure (except febrile) or increased risk of seizure. (N.B. We are not aware of evidence that LIFU can induce seizures; however, we decided to incorporate similar safeguards to those used in TMS studies.
* 6. Contraindications for MRI, including any metal in the head, metallic particles in the eye, implanted cardiac pacemaker or any intracardiac lines, implanted neurostimulators, intracranial implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or implanted medical pumps.
* 7. Subjects with significant neurological disorder or insult, ablative surgery or DBS.
* 8. History of substance abuse including alcohol use disorder within the past 6 months (except nicotine and caffeine).
* 9. Unstable medical or neurological condition
* 10. Women of childbearing potential and not using a medically accepted form of contraception such as: the consistent use of an approved hormonal contraception (birth control pill/patches, rings); an intrauterine device (IUD); Contraceptive injection (Depo-Provera); double barrier methods (diaphragm with spermicidal gel or condoms with contraceptive foam); Sexual abstinence (no sexual intercourse) or sterilization.
* 11. Taking regular dose of benzodiazepines in excess of equivalent to clonazepam 4 mg per day.
* 12. Mini-Mental State Exam (MMSE) less than 24
* 13. Current or prior history, per DSM-5 criteria, of bipolar I disorder, schizophrenia or other psychotic disorders, autism or autistic spectrum disorders, borderline PD, antisocial PD, body dysmorphic disorder, hoarding disorder (symptoms of hoarding disorder as part of the OCD diagnosis are allowed, a current diagnosis of Tourette's disorder. Co-morbid depression is allowed as long as OCD is considered primary.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Acute changes in domains of mood, anxiety, alertness in response to VS LIFU after each sonication session as assessed by the Likert scale. | 6 months
  This outcome measure will utilize the "Likert Scale" to assess the measure.This scale allows subjects to measure their mood, anxiety, and alertness by marking a scale numbered 0 through 4 with 0 being "Not at All" and 4 being "Extremely." This scale includes several items in which the subjects can indicate how they feel (Positive, negative, anxious, energetic, etc.).
Primary study endpoint for OCD severity will be change in Y-BOCS score after 6 sonication sessions compared to baseline. | 6 months
  Y-BOCS (Yale-Brown Obsessive Compulsive Scale) is a scale utilized to measure OCD. This scale includes a section in which subjects may mark "current/past" to indicate obsessions and compulsions. This scale also includes a section where subjects can indicate any obsessions or compulsions on a scale of 0 (no symptoms) to 5 (near constant symptoms).
  A reduction of 35% will be deemed a responder.
Safety and tolerability will be assessed using the frequency of subjects with serious adverse events (SAEs), AEs leading to discontinuation, and AEs judged to be related to LIFU. | 6 months
  Any AE's reported by the subject will be reviewed by the study PI to determine if an event caused harm or placed a subject/non-subject at an increased risk of harm, if the event was foreseeable, if the event is related or will impact research activities, and the specificity and severity of the event. AE's will be reported according to BCM reporting requirements.
Feasibility will be evaluated by determining the tolerability of the procedure for subjects as assessed by the Likert scale, and the technical ability of LIFU to modulate the desired target by MRI review. | 6 months
  The feasibility of this outcome measure works in tandem with Outcome 1 of "acute changes in mood, anxiety, and alertness" in that the Likert scale also allows us to determine the tolerability of the procedures based on the subject responses. Technical ability of LIFU to modulate the desired target via regional target engagement as reflected in changes in cerebral blood flow (CBF) using arterial spin labeling (ASL) perfusion MRI after stimulation as compared to baseline (CBF). Neurocircuit target engagement is also reflected in changes in effective connectivity from BOLD fMRI

CONTACTS AND LOCATIONS:
Overall Officials: Wayne Goodman, MD, Principal Investigator — Baylor College of Medicine
Locations (3):
- United States (3):
  - Massachussetts General Hospital, Boston, Massachusetts
  - Baylor College of Medicine, Houston, Texas
  - MD Anderson, Houston, Texas